CLINICAL TRIAL: NCT00994955
Title: Selective Retina Therapy (SRT) for Clinically Significant Diabetic Macular
Brief Title: Selective Retina Therapy (SRT) for Clinically Significant Diabetic Macular Edema
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Medical Laser Center Lübeck, Germany (Unknown); St Thomas (Ambiguous)
Responsible Party: Principal Investigator, Jost Hillenkamp, Oberarzt, Dept. of Ophthalmology, University of Schleswig-Holstein, Kiel, Germany, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SRT-1
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Diabetic Macular Edema
Keywords: SRT; laser; diabetic macular edema; diabetes; Clinically significant diabetic macular edema
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- selective retina therapy (SRT) (Experimental): Focal laser treatment with an SRT-Laser which selectively affects the retinal pigment epithelium while sparing the photoreceptor layer.
  Interventions: Device: selective retina therapy (SRT)

INTERVENTIONS:
Device: selective retina therapy (SRT) — laser treatment

SUMMARY:
Selective Retina Therapy (SRT) is an effective and safe laser treatment of clinically significant diabetic macular edema which targets the retinal pigment epithelium while sparing the neurosensory retina.

DETAILED DESCRIPTION:
Abstract:

OBJECTIVE: To evaluate effectivity and safety of Selective Retina Therapy (SRT) for diabetic macular edema (DME).

DESIGN: Prospective two-center interventional uncontrolled case series. PARTICIPANTS: 39 eyes of 39 patients with previously untreated non-ischemic DME.

INTERVENTION: Focal laser treatment with an SRT-Laser which selectively affects the retinal pigment epithelium while sparing the photoreceptor layer. The pulse energy was individually adjusted to achieve angiographically visible but funduscopically invisible effects. Optoacoustic measurements were performed to detect the individual threshold of RPE damage during laser treatment and correlated with funduscopy and fundus fluorescein angiography (FFA) or indocyanine green angiography. Follow-up at 3 and 6 months post treatment included best-corrected ETDRS visual acuity (BCVA), FFA, fundus photography, and retinal thickness measured by optical coherence tomography (OCT).

MAIN OUTCOME MEASURES: Change of BCVA, change of retinal thickness, presence of hard exudates and leakage in FFA, specificity and sensitivity of optoacoustic measurements.

RESULTS: Mean BCVA improved from 43.7 letters (standard deviation, SD=9.1) at baseline to 46.1 letters (SD=10.5) at 6 months follow-up (p=0.02). BCVA improved (> 5 letters) or remained stable (+/- 5 letters) in 84% of eyes. 13% of eyes improved by ≥ 10 letters while 16% of eyes lost more than 5 letters. There was no severe loss of vision (loss of ≥ 15 letters). Overall, mean central retinal thickness, hard exsudates and leakage in FFA did not change significantly (p>0.05) while improvement of BCVA correlated with a reduction of hard exsudates and central retinal thickness. Specificity and sensitivity of detecting the angiographic visible threshold of RPE damage by optoacoustic measurements were 86% and 70%, respectively. No adverse effects or pain were noted during or after treatment.

CONCLUSION: SRT is an effective and safe treatment of DME with functional and anatomical improvement or stabilization in most patients. Optoacoustic measurements are suitable to detect the individual threshold of RPE damage.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years and the presence of clinically significant DME according to the criteria of the ETDRS study

Exclusion Criteria:

* Ischemic diabetic macular edema, significant media opacity compromising the interpretation of fluorescein angiography and fundus photography, previous intraocular surgery, previous macular laser treatment, other retinal or ocular diseases, and known allergic hypersensitivity to fluorescein, indocyanine green, or iodine. General exclusion criteria included pregnancy or breast-feeding and significant medical conditions such as renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
best-corrected visual acuity | 2 years

SECONDARY OUTCOMES:
change of retinal thickness, presence of hard exudates and leakage in FFA, specificity and sensitivity of optoacoustic measurements | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jost Hillenkamp, MD, Principal Investigator — Dept. of Ophthalmology, University Medical Center Schleswig-Holstein, Kiel Campus